CLINICAL TRIAL: NCT04991311
Title: A Single-Center Phase 3b Trial Investigating the Long-term Effect on Intestinal Absorption, Nutritional Status and Long-Term Safety of Treatment With Glepaglutide in Patients With Short Bowel Syndrome (SBS)
Brief Title: The Long-term Effect on Intestinal Absorption and Safety of Treatment With Glepaglutide in Patients With Short Bowel Syndrome
Acronym: EASE SBS 4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zealand Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZP1848-20060; 2020-005194-27 (EudraCT Number); U1111-1260-2961 (Other: WHO)
Record Dates: First submitted 2021-07-14; First posted 2021-08-05 (Actual); Results first posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-09

CONDITIONS: Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- once-weekly glepaglutide (Experimental): All participants will receive 10 mg of glepaglutide as once-weekly injections under the skin (subcutaneous, s.c.)
  Interventions: Drug: Glepaglutide

INTERVENTIONS:
Drug: Glepaglutide — Glepaglutide will be delivered in a single-use autoinjector.
  Other Names: ZP1848

SUMMARY:
The purpose of this trial is to investigate the long-term effect of glepaglutide on the intestinal absorption, nutritional status of participants with Short Bowel Syndrome (SBS). The trial will also investigate whether glepaglutide is safe during long-term use. All participants in the trial will receive glepaglutide injections.

Participants will have 14 visits with the study doctor. At 2 of these, participants will spend 48 hours at the trial site, one visit at the start of the trial and one after 24 weeks of treatment with glepaglutide. At all visits, participants will meet with trial staff and will have blood tests along with other clinical checks and tests done. Participants will be asked about their health and medical history.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial
* Age greater than or equal to 18 years and less than or equal to 90 years at screening
* Stable condition of SBS either with intestinal failure (SBS-IF) or intestinal insufficiency. For patients with SBS-IF, a stable condition is defined as less than 25 percent change in parenteral support (PS) volume or energy content for 4 weeks prior to screening.
* Stable body weight (less than 5 percent change in weight in the 3 months prior to screening)
* Wet weight of fecal excretion greater than or equal to 1500 grams per day demonstrated during a hospital stay prior to screening

Exclusion Criteria:

* More than 2 SBS-related or PS-related hospitalizations (e.g., catheter-related bacteremia/sepsis, bowel obstruction, severe water-electrolytes disturbances, etc.) within 6 months prior to screening
* Poorly controlled inflammatory bowel disease (IBD) that is moderately or severely active or fistula interfering with measurements or examinations required in the trial
* Current bowel obstruction
* Known radiation enteritis or significant villous atrophy, e.g., due to active celiac disease
* Cardiac disease defined as: decompensated heart failure (New York Heart Association [NYHA] Class III-IV), unstable angina pectoris, and/or myocardial infarction within the last 6 months prior to screening
* Any history of colon cancer. History of any other cancers (except margin-free resected cutaneous basal or squamous cell carcinoma or adequately treated in situ cervical cancer) unless disease-free state for at least 5 years
* Use of glucagon-like peptide-1 (GLP-1), GLP-2, human growth hormone (HGH), somatostatin, or analogs thereof, within 3 months prior to screening

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zealand Pharma, Study Director — Zealand Pharma
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at a single site in Denmark. The study was planned to enroll a minimum of 6 and a maximum of 16 patients with SBS intestinal failure (SBS-IF) or SBS intestinal insufficiency (SBS-II). First patient recruited was on 10 Aug 2021.
Pre-assignment Details: A total of 12 patients were screened: 1 patient failed the screening, 1 patient was withdrawn before receiving investigational product.
Groups:
- Once-weekly Glepaglutide: All participants received glepaglutide 10 mg once weekly for 52 weeks as injections under the skin (subcutaneous, s.c.), with a subsequent 4-week follow up period.
  Glepaglutide: Glepaglutide was delivered in a single-use autoinjector.
Period: Overall Study
Arm/Group | Once-weekly Glepaglutide
Started | 10
Completed | 9
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Once-weekly Glepaglutide: All participants received 10 mg of glepaglutide as once-weekly injections under the skin (subcutaneous, s.c.)
  Glepaglutide: Glepaglutide was delivered in a single-use autoinjector.
Arm/Group | Once-weekly Glepaglutide
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (15.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Denmark | 10
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.1 (2.32)

OUTCOME MEASURES:

1. Primary Outcome: Change in Absorption of Wet Weight/Fluids
Description: Measured by 48-hour metabolic balance studies. The metabolic balance study measured the total intake and output of energy, macronutrients (lipids, carbohydrates, proteins) and micronutrients. The oral diet (food and fluids) was assessed by duplicate meals and liquids. During the metabolic balance study, the patients collected duplicate portions of all fluids and liquids covering 24-hour periods. Likewise, all output (ostomy output, diarrhea and urine production) was collected, quantified and analyzed.
Time Frame: from Week 0 (baseline) to Week 24
Measure: Mean (Standard Deviation); unit: g/day
Groups:
- Baseline Group - Week 0: Absorption of wet weight/fluids measured at baseline visit (Week 0).
- Week 24 Group: Absorption of wet weight/fluids measured at Week 24 visit. The group is the same as the group at Week 0 visit.
Arm/Group | Baseline Group - Week 0 | Week 24 Group
Number analyzed (Participants) | 10 | 10
g/day | 841.6 (1839.10) | 1240.0 (1529.74)
Statistical Analysis 1: Comparison: Baseline Group - Week 0 vs Week 24 Group; The participants in both comparison groups are the same; Test type: Superiority; p = 0.0585, Paired t-test (2-sided, alpha=0.05); Mean Difference (Final Values) = 398.4, 95% CI 2-sided [-17.6 to 814.4], Standard Deviation 581.6

2. Secondary Outcome: Change in Absorption of Energy
Description: Oral intake minus fecal excretion: measured by 48-hour metabolic balance studies. The metabolic balance study measured the total intake and output of energy, macronutrients (lipids, carbohydrates, proteins) and micronutrients. The oral diet (food and fluids) was assessed by duplicate meals and liquids. During the metabolic balance study, the patients collected duplicate portions of all fluids and liquids covering 24-hour periods. Likewise, all output (ostomy output, diarrhea and urine production) was collected, quantified and analyzed. Energy absorption was measured by bomb calorimetry.
Time Frame: from Week 0 (baseline) to Week 24
Measure: Mean (Standard Deviation); unit: kJ/day
Groups:
- Once-weekly Glepaglutide: All participants received glepaglutide 10 mg once weekly for 52 weeks as injections under the skin (subcutaneous, s.c.) with a subsequent 4-week follow up period.
Arm/Group | Once-weekly Glepaglutide
Number analyzed (Participants) | 10
kJ/day | 1037.7 (1182.18)

3. Secondary Outcome: Change in Absorption of Carbohydrates
Description: as for outcome 1
Time Frame: from Week 0 (baseline) to Week 24
Measure: Mean (Standard Deviation); unit: g/day
Arm/Group | Once-weekly Glepaglutide
Number analyzed (Participants) | 10
g/day | 39.8 (48.31)

4. Secondary Outcome: Change in Absorption of Lipids
Description: as for outcome 1
Time Frame: from Week 0 (baseline) to Week 24
Measure: Mean (Standard Deviation); unit: g/day
Arm/Group | Once-weekly Glepaglutide
Number analyzed (Participants) | 10
g/day | 10.5 (26.56)

5. Secondary Outcome: Change in Absorption of Proteins
Description: as for outcome 1
Time Frame: from Week 0 (baseline) to Week 24
Measure: Mean (Standard Deviation); unit: g/day
Arm/Group | Once-weekly Glepaglutide
Number analyzed (Participants) | 10
g/day | 1.0 (1.65)

6. Secondary Outcome: Change in Absorption of Sodium
Description: as for outcome 1
Time Frame: from Week 0 (baseline) to Week 24
Measure: Mean (Standard Deviation); unit: mmol/day
Arm/Group | Once-weekly Glepaglutide
Number analyzed (Participants) | 10
mmol/day | 28.0 (83.64)

7. Secondary Outcome: Change in Absorption of Potassium
Description: as for outcome 1
Time Frame: from Week 0 (baseline) to Week 24
Measure: Mean (Standard Deviation); unit: mmol/day
Arm/Group | Once-weekly Glepaglutide
Number analyzed (Participants) | 10
mmol/day | 1.9 (26.44)

8. Secondary Outcome: Change in Absorption of Calcium
Description: as for outcome 1
Time Frame: from Week 0 (baseline) to Week 24
Measure: Mean (Standard Deviation); unit: mmol/day
Arm/Group | Once-weekly Glepaglutide
Number analyzed (Participants) | 10
mmol/day | 1.3 (6.42)

9. Secondary Outcome: Change in Absorption of Magnesium
Description: as for outcome 1
Time Frame: from Week 0 (baseline) to Week 24
Measure: Mean (Standard Deviation); unit: mmol/day
Arm/Group | Once-weekly Glepaglutide
Number analyzed (Participants) | 10
mmol/day | -2.2 (5.06)

10. Secondary Outcome: Change in Weekly Parenteral Support (PS) Volume
Description: Only for participants with Short Bowel Syndrome with Intestinal Failure (SBS-IF). PS use was recorded in patient diaries throughout the trial, including type and volume used.
Time Frame: from Week 0 (baseline) to Week 12
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Once-weekly Glepaglutide
Number analyzed (Participants) | 8
mL | -4688.1 (3150.67)

11. Secondary Outcome: Change in Weekly PS Volume
Description: Only for participants with SBS-IF. PS use was recorded in patient diaries throughout the trial, including type and volume used.
Time Frame: from Week 0 (baseline) to Week 24
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Once-weekly Glepaglutide
Number analyzed (Participants) | 8
mL | -5312.6 (5463.54)

12. Secondary Outcome: Change in Weekly PS Carbohydrates
Description: as for outcome 11
Time Frame: from Week 0 (baseline) to Week 12
Measure: Mean (Standard Deviation); unit: kJ
Arm/Group | Once-weekly Glepaglutide
Number analyzed (Participants) | 8
kJ | -3547.1 (6375.32)

13. Secondary Outcome: Change in Weekly PS Carbohydrates
Description: as for outcome 11
Time Frame: from Week 0 (baseline) to Week 24
Measure: Mean (Standard Deviation); unit: kJ
Arm/Group | Once-weekly Glepaglutide
Number analyzed (Participants) | 8
kJ | -4914.8 (2452.10)

14. Secondary Outcome: Change in Weekly PS Lipids
Description: as for outcome 11
Time Frame: from Week 0 (baseline) to Week 12
Measure: Mean (Standard Deviation); unit: kJ
Arm/Group | Once-weekly Glepaglutide
Number analyzed (Participants) | 8
kJ | -260.3 (1361.60)

15. Secondary Outcome: Change in Weekly PS Lipids
Description: as for outcome 11
Time Frame: from Week 0 (baseline) to Week 24
Measure: Mean (Standard Deviation); unit: kJ
Arm/Group | Once-weekly Glepaglutide
Number analyzed (Participants) | 8
kJ | -42.2 (1869.08)

16. Secondary Outcome: Change in Weekly PS Proteins
Description: as for outcome 11
Time Frame: from Week 0 (baseline) to Week 12
Measure: Mean (Standard Deviation); unit: kJ
Arm/Group | Once-weekly Glepaglutide
Number analyzed (Participants) | 8
kJ | -879.3 (1939.60)

17. Secondary Outcome: Change in Weekly PS Proteins
Description: as for outcome 11
Time Frame: from Week 0 (baseline) to Week 24
Measure: Mean (Standard Deviation); unit: kJ
Arm/Group | Once-weekly Glepaglutide
Number analyzed (Participants) | 8
kJ | -1057.7 (983.93)

18. Secondary Outcome: Change in Weekly PS Sodium
Description: as for outcome 11
Time Frame: from Week 0 (baseline) to Week 12
Measure: Mean (Standard Deviation); unit: mmol
Arm/Group | Once-weekly Glepaglutide
Number analyzed (Participants) | 8
mmol | -473.7 (440.09)

19. Secondary Outcome: Change in Weekly PS Sodium
Description: as for outcome 11
Time Frame: from Week 0 (baseline) to Week 24
Measure: Mean (Standard Deviation); unit: mmol
Arm/Group | Once-weekly Glepaglutide
Number analyzed (Participants) | 8
mmol | -475.7 (506.37)

20. Secondary Outcome: Change in Weekly PS Potassium
Description: as for outcome 11
Time Frame: from Week 0 (baseline) to Week 12
Measure: Mean (Standard Deviation); unit: mmol
Arm/Group | Once-weekly Glepaglutide
Number analyzed (Participants) | 8
mmol | -35.6 (73.88)

21. Secondary Outcome: Change in Weekly PS Potassium
Description: as for outcome 11
Time Frame: from Week 0 (baseline) to Week 24
Measure: Mean (Standard Deviation); unit: mmol
Arm/Group | Once-weekly Glepaglutide
Number analyzed (Participants) | 8
mmol | -58.9 (51.64)

22. Secondary Outcome: Change in Weekly PS Magnesium
Description: as for outcome 11
Time Frame: from Week 0 (baseline) to Week 12
Measure: Mean (Standard Deviation); unit: mmol
Arm/Group | Once-weekly Glepaglutide
Number analyzed (Participants) | 8
mmol | 1.6 (9.02)

23. Secondary Outcome: Change in Weekly PS Magnesium
Description: as for outcome 11
Time Frame: from Week 0 (baseline) to Week 24
Measure: Mean (Standard Deviation); unit: mmol
Arm/Group | Once-weekly Glepaglutide
Number analyzed (Participants) | 8
mmol | -5.8 (14.84)

24. Secondary Outcome: Anti-glepaglutide Antibodies
Description: Monitored throughout the trial at baseline (Week 0) and weeks 4, 12, 24, 52 and 56
Time Frame: Week 56
Measure: Count of Participants; unit: Participants
Arm/Group | Once-weekly Glepaglutide
Number analyzed (Participants) | 10
Participants | 9

25. Secondary Outcome: Reactivity to ZP1848
Description: Monitored throughout the trial at baseline (Week 0) and weeks 4, 12, 24, 52 and 56. Anti-drug antibodies (ADA) positive samples were analyzed for reactivity to ZP1848.
Time Frame: Week 56
Measure: Count of Participants; unit: Participants
Arm/Group | Once-weekly Glepaglutide
Number analyzed (Participants) | 10
Participants | 8

26. Secondary Outcome: Cross-reactivity to Glucagon-like Peptide-2 (GLP-2)
Description: Monitored throughout the trial at baseline (Week 0) and weeks 4, 12, 24, 52 and 56. ADA positive samples were analyzed for cross-reactivity to glucagon-like peptide-2 (GLP-2).
Time Frame: Week 56
Measure: Count of Participants; unit: Participants
Arm/Group | Once-weekly Glepaglutide
Number analyzed (Participants) | 10
Participants | 1

27. Secondary Outcome: Glepaglutide Neutralizing Antibodies
Description: Monitored throughout the trial at baseline (Week 0) and weeks 4, 12, 24, 52 and 56
Time Frame: Week 56
Measure: Count of Participants; unit: Participants
Arm/Group | Once-weekly Glepaglutide
Number analyzed (Participants) | 10
Participants | 8

ADVERSE EVENTS:
Time Frame: Safety data cover the period since the first administrated dose till Week 56.
Arm/Group | Once-weekly Glepaglutide
All-Cause Mortality (participants affected / at risk) | 1/10
Serious Adverse Events (participants affected / at risk) | 6/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Once-weekly Glepaglutide (N=10)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Stoma obstruction (Injury, poisoning and procedural complications) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pelvic fluid collection (Gastrointestinal disorders) | 1 (3)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Device related sepsis (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Stoma site abscess (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Once-weekly Glepaglutide (N=10)
Weight decreased (Investigations) | 3 (3)
Gastrointestinal stoma output abnormal (Investigations) | 2 (2)
Urine output decreased (Investigations) | 2 (2)
Weight increased (Investigations) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Gastrointestinal stoma output increased (Investigations) | 1 (1)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 8 (10)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Hot flush (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3)
Post viral fatigue syndrome (Nervous system disorders) | 1 (1)
Injection site pain (General disorders) | 7 (129)
Injection site reaction (General disorders) | 5 (19)
Oedema peripheral (General disorders) | 5 (6)
Injection site pruritus (General disorders) | 3 (26)
Fatigue (General disorders) | 2 (2)
Injection site erythema (General disorders) | 2 (22)
Influenza like illness (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Thirst (General disorders) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal hernia (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Stomal hernia (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Torticollis (Musculoskeletal and connective tissue disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (7)
COVID-19 (Infections and infestations) | 2 (3)
Catheter site infection (Infections and infestations) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (2)
Erysipelas (Infections and infestations) | 1 (2)
Folliculitis (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (2)
Sinusitis (Infections and infestations) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (4)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1)
Stoma site dermatitis (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-07-02): https://cdn.clinicaltrials.gov/large-docs/11/NCT04991311/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT04991311/SAP_001.pdf